CLINICAL TRIAL: NCT04280679
Title: Minimally Invasive Treatment of Insufficient Superficial and Perforating Veins of the Lower Limb Using High Intensity Focused Ultrasound (HIFU) Generated by Sonovein 2: a Single Center Prospective Study
Brief Title: Treatment of Insufficient Superficial and Perforatring Veins of the Lower Limb Using HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-VN-002
Record Dates: First submitted 2020-02-11; First posted 2020-02-21 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Varicose Veins; Veins Diseases; Varicose Ulcer
Keywords: HIFU; High Intensity Focused Ultrasound
MeSH Terms: conditions — Varicose Veins; Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm of patient treated by HIFU (Other): Compression bandages
  Interventions: Device: Sonovein 2

INTERVENTIONS:
Device: Sonovein 2 — Patient are treated with the HIFU device and the pysician is doing a compressive bandage

SUMMARY:
This is a one-arm, open label, prospective, single center study to evaluate clinical standardization with Theraclion's Sonovein 2 HIFU device.

The original Sonovein device was tested in a clinical trial in 50 subjects and received CE Mark. That device has been updated yielding the current version of Sonovein 2. Based on the technical similarities between both devices in term of design, performance and principle of operation, the clinical data for Sonovein is sufficient to assure conformity of the Sonovein 2 with the respected essential requirements. At the same time, the compagny wishes to pursue the standardisation of the clinical practice with the second generation device and is, therefore, conducting this limited trial in 20 evaluable cases (from the planned 22 patients to be included). A "case" is defined as procedure conducted on a distinct vein.

DETAILED DESCRIPTION:
The Sonovein 2 system provides high intensity focused ultrasound (HIFU) abaltion of soft tissue. The energy is delievered via an extra-corporeal treatment probe, which includes an imaging system. The high energy ultrasound waves propagate through the skin and are focused on a portion of the target tissue, generating intense heat and causing local cell apoptosis and progressive tissue volume reduction over the following months in the tissue within the focal area. The process is then repeated in a stepwize fashion to destroy the targeted tissues. The Sonovein 2 system is comprised of several components, including the console, treatment arm containing the visualization and treatment unit (VTU), a computer with touchscreen user interface. In addition, the Sonovein 2 system is intended to be used in conjunction with a disposable cooling and coupling system known as ePack.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for venous procedure involving lower limb superficial insufficiency involving reflux in the segment to be treated
2. Physical condition allowing ambulation after the procedure
3. Availability of the patient for all the follow-up visits
4. Targeted tissue reachable for treatment with the device-meaning between 5mm and 26mm below the skin surface
5. Age over 18 years of age at the time of enrollment
6. No acute venous thrombosis
7. No complete, or near complete deep vein thrombosis
8. Patient has signed a written informed consent
9. Targeted structure sonographically visible

Exclusion Criteria:

1. Patient is pregnant or nursing
2. Known allergic reaction to anesthetic to be used
3. Legally incapacitated or imprisoned patients
4. Patient's vein target not clearly visible on the ultrasound images (B mode) at the inclusion visit
5. Patient participating in another clinical trial involving an investigational drug, device or biologic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Reduction of venous reflux | 3 months
  As measured by ultrasound

SECONDARY OUTCOMES:
Emergent Adverse Events | 3 months
  Measure of AEs and SAEs recorded in AE form at each visit
Measurement of the need to use tumescence anesthesia during the procedure | 3 months
  Evaluated dichotomously present/absent
Measurement of the need to use adjunctive procedure for treating the reflux | 3 months
  Evaluated dichotomously present/absent

CONTACTS AND LOCATIONS:
Overall Officials: Alfred OBERMAYER, MD, Principal Investigator — Karl Landsteiner Insitut fur funktionelle Phlebochirurgie
Locations (1):
- Karl Landsteiner Institut für funktionelle Phlebochirurgie, Melk, Austria

IPD SHARING:
Plan to Share IPD: No